CLINICAL TRIAL: NCT04781686
Title: Apatinib Plus Camrelizumab Combined With Docetaxel and S1 in First-line Treatment for Metastatic Gastric Cancer: HCCSC G05 Trial
Brief Title: Apatinib Plus Camrelizumab Combined With Docetaxel and S1 in First-line Treatment for Metastatic Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhou Fuxiang (Other)
Collaborators: Hubei Cancer Hospital (Other); Henan Provincial People's Hospital (Other); Huangshi Central Hospital (Other)
Responsible Party: Sponsor-Investigator, Zhou Fuxiang, Professor, Zhongnan Hospital
Organization: Zhongnan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCCSC G05
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Metastatic Gastric Adenocarcinoma; Metastatic Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — camrelizumab; apatinib; S 1 (combination); Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- First-line treatment (Experimental): First-line treatment: Apatinib plus Camrelizumab combined with Docetaxel and S1 for six cycles.
  Maintenance treatment: Apatinib and Camrelizumab
  Interventions: Drug: Camrelizumab; Drug: Apatinib Mesylate; Drug: S1; Drug: Docetaxel injection

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab (200mg) will be given i.v. on day 1 of each 3-week cycle
  Other Names: SHR-1210
Drug: Apatinib Mesylate — Apatinib (250mg) will be administered orally once a day .
Drug: S1 — S1 (BSA<1.25 40mg, BSA >=1.25-<1.5 50mg, BSA >=1.5 60mg) will be administered orally twice daily on days 1-7 of each 3-week cycle
Drug: Docetaxel injection — Docetaxel (75mg/m2 IV.drop) will be administered on day 1 of each 3-week cycle, for six cycles.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Apatinib plus Camrelizumab combined with docetaxel and S-1 as the first-line treatment of metastatic adenocarcinoma of gastric and gastroesophageal junction.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years;
2. Has histologically or cytologically diagnosed with unresectable locally advanced or metastatic gastric adenocarcinoma (GC) including gastroesophageal junction adenocarcinoma;
3. Human epidermal growth factor receptor 2 (HER2) negative: immunohistochemical (IHC) - or +; IHC ++ and fluorescence in situ hybridization (FISH) -;
4. No previous systemic therapy (chemotherapy, targeted therapy, immunotherapy, biological therapy, etc.) for GC/GEJ. Subjects with previous adjuvant/neo-adjuvant therapy completed more than 6 months can be enrolled. Anti-tumor traditional Chinese medicine is forbidden within 2 weeks before the first cycle chemotherapy. Patients are allowed to receive palliative radiotherapy (primary tumor or metastasis), but lesions in radiation field cannot be defined as target lesions for assessing objective response, and radiotherapy-related adverse reactions must be restored to at least grade 1；
5. Expected survival time ≥ 3 months;
6. Eastern Cooperative Group (ECOG) performance status score 0 or 1;
7. Weight ≥40kg, or BMI>18;
8. 1 measurable lesions at least should be detected by CT/MRI examination in accordance with the RECIST(Response Evaluation Criteria In Solid Tumors）1.1;
9. All acute toxic events (excluding hair loss, fatigue and hearing loss) caused by previous anti-tumor treatments or surgery are alleviated to grade 0-1 (according to NCI CTCAE version 5.0) or to the level specified by the inclusion/exclusion criteria of this study；
10. The main organ function of cases should be normal, and meet the following criteria:

    ① Absolute neutrophil count (ANC)≥1.5×109/L, platelet (PLT) ≥80×109/L;

    ② Total bilirubin (TBIL) <1.5 upper limit of normal (ULN), ALT (glutamic-pyruvic transaminase）and AST(glutamic-oxalacetic transaminase)≤2.5ULN. For subjects with liver metastases, ALT and AST≤5 ULN, serum Cr≤1.5ULN or endogenous creatinine clearance >50ml /min (Cockcroft-Gault formula);

    ③ International normalized ratio (INR) <1.5, prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 ULN;

    ④ Urine protein<2+; if urine protein≥2+, the 24-hour urine protein quantitative detection value must be ≤1g;
11. Females of childbearing potential (FOCBP), who are not surgically sterile or postmenopausal, must conduct pregnancy test (serum or urine) within 7 days before enrollment, and the results are negative, and willing to use appropriate contraception during the study period until at least 3 months after the last administration of the test drugs. Non-sterilized males who are sexually active must agree to use adequate contraception during the study period a until at least 3 months after the last administration of the test drugs;
12. Fully understand the study and voluntarily sign the informed consent form (ICF); willing and able to comply with planned visits, treatments, laboratory examinations and other procedures.

Exclusion Criteria:

1. HER2 positive cancer: IHC+++, IHC++ and FISH+;
2. Pathological classification of tumor is squamous carcinoma or undifferentiated carcinoma or other types;
3. The interval between disease progression and previous anti-tumor therapy for locally advanced is less than six months;
4. Central nervous system（CNS）metastases with clinical symptoms for example cerebral edema, spinal cord compression, cancerous meningitis, leptomeningeal disease, and/or progressive growth. For subjects with CNS metastases that have been adequately treated, and the neurological symptoms can return to baseline levels at least 2 weeks before enrollment (except for residual signs or symptoms related to treatment), can be enrolled. In addition, subjects must stop corticosteroids at least 2 weeks before enrollment;
5. Gastrointestinal bleeding that could not be effectively controlled; gastrointestinal perforation and/or gastrointestinal fistula occurred within 6 months before enrollment; arterial/venous thrombosis occurred within 6 months before enrollment, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism;
6. Pleural fluid, ascites, or pericardial effusion that could not be controlled within 7 days before enrollment;
7. Weight loss is more than 20% within 2 months before enrollment;
8. Major surgery performed within 28 days before enrollment (tissue biopsy for diagnosis and central venous catheter placement via peripheral vein are allowed). used immunosuppressive drugs within 7 days before enrollment, excluding nasal spray and inhaled corticosteroids or physiological doses of systemic steroid hormones (≤10 mg/d prednisone or equivalent other kinds of corticosteroids);
9. Other malignancy disease history within five years, with the exception of basal cell carcinoma or squamous carcinoma of skin, superficial bladder carcinoma, and carcinoma in situ (such as Intraductal carcinoma in situ of the breast, cervical cancer in situ, etc.);
10. With history of check point inhibitor treatment, for instance PD-1/PD-L1/ PD-L2/CD137/CTLA-4 antibody agent, and other drug stimulatory or co-inhibitory T-cell receptor;
11. Any active or suspected autoimmune diseases. Subjects who do not require systemic immunosuppressive therapy can be enrolled, such as type I diabetes, hypothyroidism that only requires hormone replacement therapy, and skin diseases that do not require systemic therapy (such as white scar wind, silver Scourge etc.).
12. Preexisting peripheral neuropathy >Grade 1;
13. Inability to swallow, chronic diarrhea and intestinal obstruction, or other factors that may affect the administration and absorption of the drug;
14. Has active infectious diseases, interstitial lung diseases, non-infectious pneumonia, or other systemic diseases that can not be controlled (such as diabetes, hypertension, pulmonary fibrosis, etc.);
15. Has a known history of HIV infection or AIDS. Has a known history of untreated or active hepatitis (active hepatitis B, defined as HBV-DNA>500 IU/ml; active hepatitis C, defined as HCV-RNA higher than the upper limit of the analytical method), or co-infection of HBV and HCV;
16. Hypertension (systolic blood pressure>140 mmHg or diastolic blood pressure>90 mmHg) that cannot be well controlled by antihypertensive drugs.
17. The following conditions occur within 6 months before enrollment: myocardial infarction, severe/unstable angina, NYHA grade 2 or higher cardiac insufficiency, clinically significant supraventricular or ventricular arrhythmia, and symptomatic congestion heart failure;
18. The use of antibiotics> 7 days within 2 weeks before enrollment, or unexplained fever> 38.5°C within 1 week before the treatment of this study (fever caused by tumors can be enrolled);
19. Has an allogenic tissue/solid organ transplant history;
20. Participated in any other clinical trials of drug within 4 weeks before enrollment, or less than 5 half-lives after the last study drug administrated.
21. Be allergic to the study drug or excipients; or have a severe allergic history to other monoclonal antibodies;
22. Has a known history of drug abuse;
23. Has a history or current evidence of any condition that might increase the risk of patients in the present trial, confound the results of the study, interfere with the cases' participation for the full duration of the study, or be not in the best interest of the participant to participate, in the opinion of the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-05-14 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 36 months
  PFS is defined as the time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator

SECONDARY OUTCOMES:
objective response rate (ORR) | 36 months
  Defined as percentage of participants achievingassessed complete response (CR) and partial response (PR) by the investigator according to the RECIST 1.1.
overall survival (OS) | 36 months
  OS is the time from enrollment to death due to any cause.
disease control rate (DCR) | 36 months
  DCR was defined as the percentage of participants who have a confirmed complete response（CR） or partial response（PR） or stable disease（SD） per RECIST 1.1 as assessed by investigator
adverse events (AE) | 36 months
  overall incidence of adverse events (AE); incidence of grade 3 or higher AE; incidence of severe adverse events (SAE); incidence of AEs leading to discontinuation of drug use; incidence of AEs leading to suspension of drug use.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hopital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No